CLINICAL TRIAL: NCT02301715
Title: Effects of Intranasal Oxytocin on Emotion Regulation to Stressful Interaction in Insecure Adolescents: a Study Protocol for a Double Blind Randomized Controlled Trial
Brief Title: Effects of Intranasal Oxytocin on Emotion Regulation in Adolescents
Acronym: ELOREA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: P/2013/160
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Emotion; Parent-Child Relations
Keywords: Intranasal oxytocin; Emotion regulation; Attachment
MeSH Terms: conditions — Emotional Regulation | interventions — Oxytocin; lactitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Active Comparator): 24 IU Oxytocin, 3 puffs per nostril, each with 4 IU OXT, intranasal application 45 min prior to the experiment
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): intranasal application, sodium chloride solution, 3 puffs per nostril, 45 min prior to the experiment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — OT spray will be performed by the research pharmacy at the University Regional Hospital Pharmacy of Besançon. The placebo contained all inactive ingredients except for the neuropeptide. Placebo and OT spray containers will be prepared to look identical and will be counterbalance to be randomly assigned by the pharmacy as well. Double blinding and randomization of patients in the two groups will also be carried out by the pharmacy service. Researchers, as well as participants, will be blinded to the content of the spray. Participants will be instructed to sit and take one puff every 30 seconds, alternating nostrils. Participant will take each dose in front of the clinician to assure correct administration and tolerability.
  Other Names: Syntocinon-Spray, Novartis
  Arms: Oxytocin
Drug: Placebo — The placebo contained all inactive ingredients except for the neuropeptide. Participants will be instructed to sit and take one puff every 30 seconds, alternating nostrils. Participant will take each dose in front of the clinician to assure correct administration and tolerability.
  Other Names: Pl
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of intranasal administration of OT on behavior and discourse of insecure adolescents during a disagreement (stressful situation) with parents.

DETAILED DESCRIPTION:
Emotional dysregulation and impaired attachment in adolescence are seen by clinical researchers as potential contributors to development of psychopathology. Recent evidence suggests that administration of intranasal OT may facilitate social interaction by attenuating the stress response to interpersonal conflict. However, to date there have been no studies investigating the effects of intranasal OT on parent-adolescent interaction and on neurophysiological emotional strategies in adolescence. To understand these mechanisms, this study examines the effects of OT on interpersonal emotional regulation in adolescent-parent stressful interaction, and on individual visual and physiological strategies in the visualizing attachment-related emotions pictures.

The main objective will be to evaluate the effect of intranasal administration of OT on behavior and discourse of insecure adolescents during a disagreement (stressful situation) with one of his parents.

Secondary is determine the effect of OT on visual exploration strategies and on the physiological responses (heart rate, galvanic skin response) on images elicited attachment-related emotions in insecure adolescents.

In this randomized, double-blind, placebo-controlled, parallel designs, 60 healthy male adolescents classified with an insecure attachment will receive 24 IU of intranasal OT or placebo, 45 min before the experimental tasks. Adolescent will be invited with his/her parent to an experimental conflict discussion. The conflict session will be videotaped and coded for verbal and nonverbal interaction behavior (e.g., eye contact, nonverbal positive/negative behavior, and self-disclosure) with GPACS. Eye tracking and physiological responses will be recorded simultaneously and continuously during pictures viewing.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of insecure attachment according to the Attachment Scale Interview
* Male adolescents (and parents) enrolled in high school or college
* Not hospitalized
* Without current or past history of neurological or psychiatric illness, including substance abuse or dependence
* Aged from 13 to 20 years
* Speaking French
* Have signed informed consent
* Affiliation to a French social security

Exclusion Criteria:

* Females
* Intellectual deficit
* Severe neurological symptoms
* Known allergies to oxytocin or to preservatives in the nasal spray
* Not speaking French
* Visual disturbances
* Chronic disease (liver failure, kidney failure, cardiovascular disease)
* Antihypertensive therapy

Ages: 13 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04-29 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Conflict discussion | 3 years
  Adolescent will be invited with his/her parent to an experimental conflict discussion. The conflict session will be videotaped and coded for verbal and nonverbal interaction behavior (e.g., eye contact, nonverbal positive/negative behavior, and self-disclosure) with GPACS.Behavioral data will be collected during each of the study visits. Drug effect will be determined by comparing data obtained during placebo and oxytocin visits.

SECONDARY OUTCOMES:
Visual patterns | 3 years
  Adolescent's eye tracking (i.e., time (ms) and frequency of fixations in an AOI) and physiological (Amplitude of SCL (microsiemens), Amplitude of SCRs (microsiemens), Time of latency (s)) responses will be recorded simultaneously and continuously during pictures viewing.

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane Vulliez-Coady, PhD, Principal Investigator — CHU Besançon
Locations (1):
- University Regional Hospital, Besançon, Franche-Comté, France